CLINICAL TRIAL: NCT06628193
Title: Study of Low-intensity Focused Ultrasound Effects on Human Memory
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Virginia Polytechnic Institute and State University (Other)
Responsible Party: Principal Investigator, Wynn Legon, Assistant Professor, Virginia Polytechnic Institute and State University
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Other
Other Study IDs: 24-999
Record Dates: First submitted 2024-09-23; First posted 2024-10-04 (Actual); Last update posted 2025-02-17 (Actual); Status verified 2025-02

CONDITIONS: Memory
Keywords: LIFU

STUDY DESIGN:
Intervention Model Description: sham-controlled, repeated measures design conducted across eight sessions
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (8):
- Sham LIFU (Sham Comparator): Sham LIFU stimulation visit with memory tasks and neuropsychological assessments.
  Interventions: Device: Sham (No Treatment)
- LIFU 1 (Experimental): LIFU stimulation with parameter set 1 visit with memory tasks and neuropsychological assessments.
  Interventions: Device: Low intensity focused ultrasound
- LIFU 2 (Experimental): LIFU stimulation with parameter set 2 visit with memory tasks and neuropsychological assessments.
  Interventions: Device: Low intensity focused ultrasound
- LIFU 3 (Experimental): LIFU stimulation with parameter set 3 visit with memory tasks and neuropsychological assessments.
  Interventions: Device: Low intensity focused ultrasound
- LIFU 4 (Experimental): LIFU stimulation with parameter set 4 visit with memory tasks and neuropsychological assessments.
  Interventions: Device: Low intensity focused ultrasound
- LIFU 5 (Experimental): LIFU stimulation with parameter set 5 visit with memory tasks and neuropsychological assessments.
  Interventions: Device: Low intensity focused ultrasound
- LIFU 6 (Experimental): LIFU stimulation with parameter set 6 visit with memory tasks and neuropsychological assessments.
  Interventions: Device: Low intensity focused ultrasound
- LIFU 7 (Experimental): LIFU stimulation with parameter set 7 visit with memory tasks and neuropsychological assessments.
  Interventions: Device: Low intensity focused ultrasound

INTERVENTIONS:
Device: Low intensity focused ultrasound — low-intensity focused ultrasound for neuromodulation applied to the head.
  Arms: LIFU 1; LIFU 2; LIFU 3; LIFU 4; LIFU 5; LIFU 6; LIFU 7
Device: Sham (No Treatment) — Sham LIFU application
  Arms: Sham LIFU

SUMMARY:
This research project is examining the effects of noninvasive brain stimulation on human memory. This study will help to better understand noninvasive brain stimulation techniques that may have the potential to aid in memory dysfunction. Subjects will undergo a magnetic resonance imaging (MRI) and a computed tomography (CT) scan, to take pictures of their brain and skull. They will receive noninvasive brain stimulation using low-intensity focused ultrasound (LIFU) sound waves, to temporarily change brain activity. Their brain signals (MRI or EEG) will be monitored to measure changes in their brain signals. Their heart rate, blood pressure, respiratory rate, eye movement and skin moisture will be monitored as well. They will complete neuropsychological batteries and memory tasks. They will complete questionnaires.

DETAILED DESCRIPTION:
This study employs a two-arm, sham-controlled, repeated measures design conducted across eight sessions:

Overall Structure

* Session 1: Baseline Assessment and Imaging
* Session 2-8: LIFU Stimulation *The order of Sessions 2-8 is ideally randomized to control for order effects. The study design allows for flexibility to accommodate varying levels of participant completion while maintaining scientific validity.

Detailed Session Breakdown Session 1: Baseline Assessment and Imaging

* Structural & Functional imaging: MRI and CT anatomical scans
* Administration of questionnaire battery Session 2-8: LIFU Stimulation or Sham
* Memory task performance
* Neuropsychological battery administration
* EEG recording
* Collection of physiological measures (HR, BP, RR, and EDR)

Design Considerations: There will be at least one week between Session 1 and Session 2, and at least 48 hours between each subsequent session. This design allows for within-subject comparisons across stimulation conditions, as well as between-subject comparisons if the full protocol is completed. The study protocol is designed to accommodate potential variability in participant availability. While full completion of all sessions is ideal, partial completion can still yield valuable data.

ELIGIBILITY:
Inclusion Criteria:

* Subjects of all ethnicities, who understand and speak English.

Exclusion Criteria:

* The exclusion criteria below are regularly implemented in MRI, CT, and EEG experiments for the safety of the subjects and for data quality assurance.

  1. Claustrophobia (scanning environment may be uncomfortable).
  2. Contraindications to MRI: including pacemaker, aneurysm clips, neurostimulators, cochlear implants, metal in eyes, steel worker, or other implants.
  3. Contraindications to CT: pregnancy
  4. Active medical disorder or treatment with potential CNS effects (e.g. Alzheimer's)
  5. History of neurologic disorder. (e.g. Parkinson's, Epilepsy, or Essential Tremor)
  6. History of head injury resulting in loss of consciousness for >10 minutes.
  7. History of alcohol or drug dependence (through self-report).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2024-11-18 (Actual); Primary Completion 2026-11 (Estimated); Study Completion 2027-05 (Estimated)

PRIMARY OUTCOMES:
Memory Task Accuracy | up to 6 weeks
  The percentage of correct responses during memory recall tasks, measured as a percentage. This metric will evaluate accuracy following LIFU stimulation compared to sham stimulation.
Memory Task Reaction Time | up to 6 weeks
  Reaction time during memory recall tasks, measured in milliseconds. This metric will assess the speed of memory recall following LIFU stimulation compared to sham stimulation.

SECONDARY OUTCOMES:
Electroencephalography(EEG) Power Spectral Analysis in Targeted Brain Regions | up to 6 weeks
  Change in theta power (4 - 8 HZ) and gamma power (30 - 100 HZ) measured by up to 64-channel EEG systems within targeted brain regions, measured in microvolts squared (uV2). This outcome will assess alterations in brain electrical activities during memory tasks.
Phase-Amplitude Coupling (PAC) Index | up to 6 weeks
  Change in the strength of phase-amplitude coupling between theta and gamma oscillations measured by up to 64-channel electroencephalography (EEG) systems, expressed as a coupling index (unitless ration). This outcome will provide insights into neural connectivity alterations during memory tasks.
Executive Function Score | up to 6 weeks
  Executive function will be assessed using standardized tools form NIH Toolbox Cognitive Battery, with results expressed as T-scores.
Attention Score | up to 6 weeks
  Attention will be measured through the NIH Toolbox Cognitive Battery, with results provided in T-scores
Processing Speed Score | up to 6 weeks
  Processing speed will be evaluated using the NIH Toolbox Cognitive Battery with scores expressed as T-scores.

CONTACTS AND LOCATIONS:
Locations (1):
- Fralin Biomedical Research Institute at VTC, Roanoke, Virginia, United States

IPD SHARING:
Plan to Share IPD: Undecided